CLINICAL TRIAL: NCT03091634
Title: The Efficacy and Safety of the Xue-Fu-Zhu-Yu Capsule in Treating qi Stagnation and Blood Stasis Syndrome: a Multicenter, Double-blind, Randomized and Placebo-controlled Trial
Brief Title: The Efficacy and Safety of the Xue-Fu-Zhu-Yu Capsule in Treatment of Qi Stagnation and Blood Stasis Syndrome.
Acronym: TROTEASOTXZC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: China Food and Drug Administration (Other Government); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hao-qiang He, master degree candidate, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HHe
Record Dates: First submitted 2017-03-17; First posted 2017-03-27 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Qi Stagnation and Blood Stasis Syndrome
Keywords: Xue-Fu-Zhu-Yu Capsule; Qi Stagnation and Blood Stasis syndrome; National Center for Complementary and Integrative Health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): the patients in this group take 6 xue-fu-zhu-yu capsules once, twice a day, for 7weeks.
  Interventions: Drug: xue-fu-zhu-yu capsule
- control group (Placebo Comparator): the patients in this group take 6 xue-fu-zhu-yu capsule simulated agents once, twice a day, for 7weeks..
  Interventions: Drug: xue-fu-zhu-yu capsule simulated agent

INTERVENTIONS:
Drug: xue-fu-zhu-yu capsule — participants are given to 6 xue-fu-zhu-yu capsule per time, twice a day. The duration is 7 weeks
  Other Names: xue fu zhu yu capsule
  Arms: test group
Drug: xue-fu-zhu-yu capsule simulated agent — participants are given to 6 xue-fu-zhu-yu capsule simulated agent per time, twice a day. The duration is 7 weeks
  Other Names: simulated agent
  Arms: control group

SUMMARY:
This is a multicenter, double-blind, randomized and placebo-controlled trial. The study aims to evaluate the effectiveness and safety of Xue-Fu-Zhu-Yu Capsule (XFZYC) for Qi Stagnation and Blood Stasis syndrome (QS&BSS). QS&BSS is one of the common Zhengs in Traditional Chinese Medicine, which manifests as various symptoms and signs, such as distending pain or tingling sensation in a fixed position, irritability or depression, dim complexion, lumps in body, blood spot under the skin, unsmooth or string-like pulse, purplish tongue or petechia in the tongue, etc. In fact, Qi stagnation and blood stasis are common pathological conditions that would occur on human body for several times in the long period of human's life. Besides, QS&BSS is associated with over 50 kinds of diseases including Coronary Heart Disease, hypertension, cerebral infarction, gastritis, arthritis, dysmenorrhea, chronic pelvic infection, skin disease, and cancer. Xue-Fu-Zhu-Yu Capsule, one of Chinese herbal medicine drugs, could perform the function of promoting Qi and activating blood to relieve the symptoms of QS&BSS, which was approved by the China Food and Drug Administration in 2002. It has been applied for QS&BSS since it was recorded in the book Correction on Errors in Medical Classics 200 years ago. In recent years, a number of clinical trials have focused on the effectiveness and safety of XFZYC on patients with QS&BSS subtype of coronary heart disease, hyperlipidemia, ischemic cerebrovascular disease, gastritis, dysmenorrhea, and arthritis in terms of the outcomes of relevant diseases. Our research group plan this randomized controlled trial to evaluate the effectiveness and safety of Xue-Fu-Zhu-Yu Capsule (XFZYC). A total of 120 patients will be enrolled at the following three hospitals: (1)Guang'anmen Hospital, China Academy of Chinese Medical Sciences, (2)Huguosi TCM Hospital Affiliated to Beijing University of Chinese Medicine, (3)Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing, China. All participants, with different kinds of disease, will receive the standard medical care according to the guidelines. Participants will undergo a 7-week treatment. The primary outcome is the total score of the Traditional Chinese Medicine Patient Reported Outcome (PRO) Scale in Patients of QS&BSS; the secondary outcome is the score of the single symptom and sign scale of QS&BSS and the score of the pain scale of QS&BSS on the day of enrollment, and at 2nd, 4th, 6th, 7th weeks. Safety outcomes include physical examination (temperature, respiration, heart rate, blood pressure, height and weight); electrocardiogram (ECG); complete blood cell count; coagulation function (prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT), fibrinogen (FIB), D-Dimer, INR); urinalysis; fecal occult blood test; Liver function (ALT, aspartate aminotransferase (AST), alkaline phosphatase (ALP), serum total bilirubin (STB), and γ-glutamyl transpeptidase (γ-GT)); renal function (Creatinine (Cr), blood urea nitrogen (BUN), and urine N-acetyl-β glucosaminidase) on the day of enrollment, and at 7th weeks.

ELIGIBILITY:
Inclusion Criteria:

* The participants diagnosed as QS&BSS;
* The age of participants is from 18 to 65;
* Participants who voluntarily signed informed consent.

Exclusion Criteria:

* Participants with other obvious Chinese medicine syndrome
* Participants diagnosed as acute myocardiac infarction, acute phase of cerebral infarction, aortic dissection and other critically illness;
* Participants with poor control of hypertension (systolic pressure >160 millimeters of mercury (mmHg) or diastolic blood pressure >100mmHg), severe heart failure and severe arrhythmia (atrial fibrillation, atrial flutter, ventricular tachycardia, paroxysmal II type II atrioventricular block and complete bundle branch block);
* Participants with severe primary diseases of heart, brain, liver, kidney and hematopoietic system, or liver function ALT or AST value >1.5 times of the upper limit of the normal value, or abnormal renal function;
* Depression or anxiety disorders participants;
* Pregnant or lactating women;
* Participants with nerve or mental illness, or unwilling to cooperate participants;
* Participants have performed a surgery in the past 4 weeks;
* Participants with the tendency of bleeding or abnormal value of disseminated intravascular coagulation (DIC) or International standard ratio (INR) or thrombocytopenia patients;
* Participants have joined in other trial in the past 1 month;
* Participants allergic to the test drug, or people with allergic constitution;
* Participants with aphasia which affects data collection.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-05-06 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The Traditional Chinese Medicine PRO Scale | baseline, 2nd,4th,6th and 7th week
  The Traditional Chinese Medicine PRO scale includes physiological domain,psychological domain,independence and social domain. And the change of the total score of the Traditional Chinese Medicine PRO Scale in Patients of QS&BSS will be assessed.

SECONDARY OUTCOMES:
The single symptom and sign scale of QS&BSS | baseline, 2nd,4th,6th and 7th week
  Patients' single symptom and sign evaluation will use the score of the single symptom and sign scale of QS&BSS. According to the degree of symptom and sign, the score is given as no = 0; mild = 1; moderate = 2; severe = 3
The pain scale of QS&BSS | baseline, 2nd,4th,6th and 7th week
  The pain will be assessed by the score of the pain scale of QS&BSS. The total score includes visual analogue scale pain index and the score of degree, duration, and frequency of pain . The position of pain will be counted independently.

OTHER OUTCOMES:
safety outcome | baseline and 7th week
  physical examination (temperature, respiration, heart rate, blood pressure, height and weight), complete blood cell count, urinalysis, stool examination, fecal occult blood test, liver function (ALT, AST, alkaline phosphatase (ALP), serum total bilirubin (STB), and γ-glutamyl transpeptidase (γ-GT)), renal function (Cr, BUN, and urine N-acetyl-β-glucosaminidase) and electrocardiogram (ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, professor, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences; Yu Liu, master, Principal Investigator — Huguosi TCM Hospital Affiliated to Beijing University of CM; Chenhao Zhang, professor, Principal Investigator — Wangjing Hospital, China Academy of Chinese Medical Sciences; Yongyan Wang, professor, Study Chair — Institute of Basic Research in Clinical Medicine; Jianyuan Tang, Study Director — China Food and Drug Administration
Locations (3):
- China (3):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing
  - Huguosi TCM Hospital Affiliated to Beijing University of CM, Beijing
  - Wangjing Hospital, China Academy of Chinese Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] He H, Chen G, Gao J, Liu Y, Zhang C, Liu C, Li H, He Q, Li J, Wang J. Xue-Fu-Zhu-Yu capsule in the treatment of qi stagnation and blood stasis syndrome: a study protocol for a randomised controlled pilot and feasibility trial. Trials. 2018 Sep 21;19(1):515. doi: 10.1186/s13063-018-2908-9. PMID 30241562